CLINICAL TRIAL: NCT00358644
Title: A Phase II Study of Decitabine For the Front-line Treatment of Older Patients With Acute Myeloid Leukemia
Brief Title: Study of Decitabine for Treatment of Older Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACO-017; NCT00238095 (obsolete NCT alias)
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2010-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Decitabine; Dacogen; MGI PHARMA, INC.
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — 20 mg/m^2, IV on days 1-5 of each 28 day cycle; until death, progression or unacceptable toxicity develops.
  Other Names: Dacogen

SUMMARY:
The purpose of this study is to estimate the rate of complete remission, as well as overall survival, in older patients with Acute Myeloid Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of AML or transformed from myelodysplastic syndrome (MDS) within 2 weeks of study enrollment.
2. Ineligible to receive intensive chemotherapy for their disease.
3. Have not received any chemotherapy within 4 weeks of study enrollment and must have recovered from any treatment-related toxicities.

Exclusion Criteria:

1. Received previous treatment for AML.
2. Previously received Vidaza.
3. Received any other investigational agents within 30 days of first dose of study drug.
4. Uncontrolled intercurrent illness.
5. Had radiotherapy within 14 days prior to study enrollment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-03; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai US Medical Services, Study Director — Eisai Inc.
Locations (3):
- United States (3):
  - Duarte, California
  - Los Angeles, California
  - St Louis, Missouri

REFERENCES:
- See also: Official website of MGI PHARMA, Inc. — http://www.mgipharma.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine 20 mg/m2 Intravenous: Decitabine 20 mg/m2 Intravenous on Days 1-5 of each 28 day cycle
Period: Overall Study
Arm/Group | Decitabine 20 mg/m2 Intravenous
Started | 55
Completed | 5
Not Completed | 50
Not completed — Progressive Disease | 21
Not completed — Adverse Event | 7
Not completed — Death | 11
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 6
Not completed — Patient not eligible for study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine 20 mg/m2 Intravenous
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 73.0 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Complete Response = Morphologic Complete Remission (mCR)
Time Frame: 1 year
Population: Intent-to-Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Decitabine 20 mg/m2 Intravenous
Number analyzed (Participants) | 55
Participants | 13
Statistical Analysis 1: Comparison: Decitabine 20 mg/m2 Intravenous; Test type: Superiority or Other; Percentage of Participants = 23.6, 95% CI [13.2 to 37.0]

ADVERSE EVENTS:
Arm/Group | Decitabine 20 mg/m2 Intravenous
Serious Adverse Events (participants affected / at risk) | 40/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine 20 mg/m2 Intravenous (N=55)
Anemia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 13
Neutropenia (Blood and lymphatic system disorders) | 4
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Blood and lymphatic system disorders) | 2
Myocardial Infarction (Cardiac disorders) | 1
Caecitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Catheter Thrombosis (General disorders) | 1
Chest Pain (General disorders) | 1
Disease Progression (General disorders) | 9
Mucosal Inflammation (General disorders) | 1
Performance Status Decreased (General disorders) | 3
Pyrexia (General disorders) | 4
Cholecystitis Acute (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Alpha Haemolytic Streptococcal Infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 6
Catheter Site Infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Clostridium Difficile Colitis (Infections and infestations) | 4
Enterocolitis Infectious (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Fungal Sepsis (Infections and infestations) | 1
Gingival Infection (Infections and infestations) | 1
Groin Abscess (Infections and infestations) | 1
Lobar Pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia Fungal (Infections and infestations) | 1
Pneumonia Klebsiella (Infections and infestations) | 1
Pneumonia Primary Atypical (Infections and infestations) | 1
Pseudomonal Bacteraemia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 8
Staphylococcal Bacteraemia (Infections and infestations) | 3
Staphylococcal Infection (Infections and infestations) | 1
Staphylococcal Sepsis (Infections and infestations) | 1
Streptococcal Bacteraemia (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 4
Urosepsis (Infections and infestations) | 1
Haemolytic Transfusion Reaction (Injury, poisoning and procedural complications) | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1
Blood Creatinine Increased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage Intracranial (Nervous system disorders) | 1
Mental Status Changes (Psychiatric disorders) | 2
Renal Failure (Renal and urinary disorders) | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine 20 mg/m2 Intravenous (N=55)
Anaemia (Blood and lymphatic system disorders) | 14
Febrile Neutropenia (Blood and lymphatic system disorders) | 17
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Atrial Fibrillation (Cardiac disorders) | 4
Sinus Tachycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 5
Ear Pain (Ear and labyrinth disorders) | 3
Conjuntival Haemorrhage (Eye disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 23
Diarrhea (Gastrointestinal disorders) | 22
Gingival Bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 28
Oral Pain (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 17
Catheter Site Pain (General disorders) | 3
Chills (General disorders) | 13
Disease Progression (General disorders) | 9
Fatigue (General disorders) | 37
Mucosal Inflammation (General disorders) | 11
Oedema (General disorders) | 11
Oedema Peripheral (General disorders) | 20
Pain (General disorders) | 10
Performance Status Decreased (General disorders) | 5
Pyrexia (General disorders) | 24
Hyperbilirubinemia (Hepatobiliary disorders) | 3
Bacteraemia (Infections and infestations) | 7
Candidiasis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 3
Clostridium Difficile Colitis (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 9
Sepsis (Infections and infestations) | 8
Staphylococcal Bacteraemia (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 8
Procedural Pain (Injury, poisoning and procedural complications) | 8
Alanine Aminotransferase Increased (Investigations) | 4
Blood Alkaline Phosphatase Increased (Investigations) | 4
Blood Creatinine Increased (Investigations) | 6
International Normalised Ratio Increased (Investigations) | 6
Weight Decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 9
Decreased Appetite (Metabolism and nutrition disorders) | 9
Fluid Overload (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 15
Headache (Nervous system disorders) | 13
Hypoaesthesia (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 10
Renal Failure (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 10
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Night Sweats (Skin and subcutaneous tissue disorders) | 5
Petechiae (Skin and subcutaneous tissue disorders) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 8
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No